CLINICAL TRIAL: NCT00120367
Title: Early Intensification of Combination Antiretroviral Therapy Including FUZEON® in the Treatment of Progressive Multifocal Leucoencephalopathy During HIV-1 Infection ANRS 125 Trial
Brief Title: Early Intensification of Antiretroviral Therapy Including Enfuvirtide in HIV-1-Related Progressive Multifocal Leucoencephalopathy (ANRS125)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-000424-16; ANRS 125
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Leukoencephalopathy, Progressive Multifocal; HIV Infections
Keywords: Leukoencephalopathy, Progressive Multifocal; HIV infections; HIV Fusion Inhibitors
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal; HIV Infections | interventions — Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide
Drug: Tenofovir-Emtricitabine

SUMMARY:
Progressive multifocal leucoencephalopathy (PML) is a rare infectious disease of the brain, provoked by the JC virus. It usually occurs in subjects with impaired immune system as during HIV infection. To date, there is no specific antiviral treatment susceptible to cure PML. But it was shown in the setting of HIV-related PML, that combination antiretroviral therapy allows a restoration of the immune system and then might stop the progression of PML.

The objective of this study is to appreciate the supplementary efficiency brought by an association of more powerful antiretroviral molecules including enfuvirtide on the evolution of PML. This research program will involve 30 patients in several centres in France. All the patients who will participate will receive enfuvirtide during 6 months in association with a combination of two or more potent antiretroviral drugs. The total duration of follow-up for a patient will be of 1 year.

DETAILED DESCRIPTION:
The aim of this open-label multicentre study is to estimate the effect of an early therapy intensification based on potent antiretroviral combination including enfuvirtide(FUZEON®) on survival in patients with HIV-1-related progressive multifocal leucoencephalopathy (PML).

To demonstrate that the observed rate is significantly superior to 45%, the inclusion of 24 patients is necessary. At last, 30 patients will be recruited towards the risk estimated at 25% of invalid inclusion.

Patients will be included on the following criteria : HIV-1 documented by Western Blot, clinical and radiological (MRI) evidence of active LEMP with clinical evolution (or deterioration) for less than 90 days, documentation of PML diagnosis for less than 30 days at the inclusion, informed consent (patient or confidence surrogate if decision making incapacity). Exclusion criteria will be the following: age less than 18-year-old ; concomitant opportunistic infection of the central nervous system; pregnancy - feeding; co-infection by the HIV2; history of immunotherapy (interleukin 2, alpha-interferon) or of treatment by FUZEON®; history of treatment by cidofovir; contra-indication to receive FUZEON ®.

An independent committee will meet regularly to estimate the validity of PML diagnosis in included patients.

The duration of the treatment by FUZEON® is 6 months in association with a combination of two or more antiretroviral molecules which will be pursued during the next 6 months. These molecules will be chosen according to the past treatment of the patients. A combination including efavirenz, lopinavir/ritonavir, and tenofovir/emtricitabine (under the shape of TRUVADA®) will be proposed to the naïve patients. For the pretreated patient(approximately a quarter of the inclusions), antiretroviral therapy will be chosen in every case on the basis of the therapeutic history and of the viral genotypes of resistance. Such association will contain at least two antiretroviral molecules, issued from two different families among the three following ones (nucleoside inhibitors of the reverse transcriptase, non-nucleoside inhibitors of the reverse transcriptase, protease inhibitors).

The projected duration of the period of inclusion will be 18 months. A total duration of 2.5 years is projected.

Evaluation criteria of the ANRS 125 trial are the following. Clinical: rate of survival and functional score (Modified Rankin Outcome Scale) to M12. Virological: evolution of the JC viral load in the CSF ; and percentage of patients with JC virus clearance of the CSF to M3 and M6. Immunological: evolution of T CD4 and T CD8 subpopulations. Evolution of the anti-JC virus specific T cell (CD4 and CD8) responses. Pharmacological: dosage of the concentration of enfuvirtide in the CSF compared with the plasma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Have confirmed laboratory diagnosis of HIV infection
* Presenting with a clinical history of active PML evolving (or continuing to deteriorate) for less than 90 days
* Diagnosis of PML documented for less than 30 days at the inclusion by cerebral imaging (MRI) AND the absence of another demonstrated etiology AND the detection of JCV DNA in the CSF by qualitative PCR.
* Signed written inform consent

Exclusion Criteria:

* Concomitant opportunistic infection of the central nervous system
* Pregnancy, breast-feeding
* Co-infection by the HIV2
* History of immunotherapy including interleukin-2 and alpha-interferon
* History of treatment by FUZEON® or by cidofovir
* Contra-indication to receive FUZEON

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Estimation by the method of Kaplan-Meier of the rate of survival at M12

SECONDARY OUTCOMES:
Rate of survival and functional score (Modified Rankin Outcome Scale) at M12
Evolution of the JC viral load in the CSF and percentage of patients with JC virus clearance of the CSF to M3 and M6
Evolution of the CD4 and CD8 T cells sub-populations and of the antivirus JC specific T cell responses at M12
Dosage of the concentration of enfuvirtide in the CSF

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Gasnault, MD, Principal Investigator — Hopital Bicetre Kremlin Bicetre France; Dominique Costagliola, Study Chair — Inserm U720
Locations (1):
- Service de Medecine interne et Maladies Infectieuses, Hopital Bicetre, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Gasnault J, Costagliola D, Hendel-Chavez H, Dulioust A, Pakianather S, Mazet AA, de Goer de Herve MG, Lancar R, Lascaux AS, Porte L, Delfraissy JF, Taoufik Y; ANRS 125 Trial Team. Improved survival of HIV-1-infected patients with progressive multifocal leukoencephalopathy receiving early 5-drug combination antiretroviral therapy. PLoS One. 2011;6(6):e20967. doi: 10.1371/journal.pone.0020967. Epub 2011 Jun 30. PMID 21738597